CLINICAL TRIAL: NCT05839769
Title: Evaluation of Carpal Tunnel Syndrome in Pregnancy
Status: Completed | Type: Observational
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, fatih sahin, MD / Principal Investigator, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Other Study IDs: 88
Record Dates: First submitted 2023-04-18; First posted 2023-05-03 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Carpal Tunnel; Carpal Tunnel Syndrome
Keywords: pregnancy; carpal tunnel syndrome
MeSH Terms: conditions — Median Neuropathy; Carpal Tunnel Syndrome | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- carpal tunnel syndrome in third trimester pregnant women: pregnant women who has CTS
  Interventions: Diagnostic Test: Evaluation of median nerve with ultrasound
- healthy pregnant women in third trimester
  Interventions: Diagnostic Test: Evaluation of median nerve with ultrasound

INTERVENTIONS:
Diagnostic Test: Evaluation of median nerve with ultrasound — ultrasound examination wrist

SUMMARY:
Carpal tunnel syndrome (CTS) is a condition that happens when the median nerve in the wrist gets compressed, causing pain, numbness, and tingling in the hand and fingers. It's a common condition that affects between 3% and 6% of people in the general population.

During pregnancy, CTS can be a bigger problem because hormonal changes can cause swelling and put more pressure on the median nerve. Studies show that CTS can affect up to 45% of pregnant women, making it important to identify and manage.

CTS can be diagnosed through a physical exam by a doctor, who will check for symptoms like pain, tingling, or weakness in the hand and fingers. Ultrasound can also be used to diagnose CTS by measuring the size of the median nerve in the wrist. This is a non-invasive imaging technique that is generally considered reliable for diagnosing CTS.

In previous studies, ultrasound has been used to measure the size of the median nerve in pregnant women with carpal tunnel syndrome (CTS). However, a new ratio of median nerve cross-sectional area to flexor carpi radialis cross-sectional area (MN-CSA/FCR-CSA) has not been studied in pregnant women. This ratio may be a more sensitive diagnostic tool for CTS because it is not affected by swelling, which is a common symptom during pregnancy that can affect the size of the median nerve.

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is a condition that arises due to the compression of the median nerve in the carpal tunnel of the wrist. The prevalence of CTS in the general population is estimated to be between 3% and 6%, with higher rates in certain occupations or activities that involve repetitive hand movements or vibrations.

During pregnancy, CTS can be particularly important due to hormonal changes that can cause an increase in fluid retention and pressure on the median nerve. The prevalence of CTS during pregnancy varies widely in the literature, with some studies reporting rates as high as 45%.

Ultrasound is a non-invasive imaging technique that can be used to diagnose CTS by measuring the cross-sectional area of the median nerve. While there is some debate regarding the normative values of median nerve cross-sectional area, ultrasound is generally considered a reliable diagnostic tool for CTS.

Previous research has utilized ultrasound to measure the cross-sectional area of the median nerve (MN-CSA) in pregnant women diagnosed with carpal tunnel syndrome (CTS). However, the potential diagnostic value of the MN-CSA/flexor carpi radialis cross-sectional area (FCR-CSA) ratio has not been examined in this population. Given that edema, a common symptom of pregnancy, may affect MN-CSA but not MN-CSA/FCR-CSA ratio, this novel ultrasound parameter may offer superior sensitivity for diagnosing CTS in pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* have undergone provocation tests during physical examination that match the median nerve distribution, and are experiencing symptoms of numbness, tingling, weakness and pain in the hands that have persisted for at least one month, and have been diagnosed with carpal tunnel syndrome through electromyography.

Exclusion Criteria:

* a history of carpal tunnel surgery
* gestational diabetes mellitus
* eclampsia or preeclampsia
* thyroid disorders
* arthropathies, hand or wrist trauma
* bilateral fractures
* atrial fibrillation
* cervical radiculopathy
* peripheral neuropathy
* thoracic outlet syndrome
* diabetes mellitus
* hypothyroidism
* hyperthyroidism
* rheumatologic disease.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant woman
Study Population: CTS in pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-09-10 (Actual)

PRIMARY OUTCOMES:
Ultrasound imaging of wrists | The prospectively designed study will conclude upon reaching a sample size of 60 participants in the third trimester of pregnancy within a 3-month period
  Ultrasonographic measurement of the 'Nerve/Tendon Ratio' (NTR) in CTS

SECONDARY OUTCOMES:
Boston Carpal Tunnel Syndrome Questionnaire | Patients were evaluated third trimester and 1 month after the birth
  The questionnaire used in this study comprises of two parts, namely the Boston Symptom Severity Scale (BSSS) and the Boston Functional Capacity Scale (BFCS). The BSSS contains 11 questions related to symptom severity, with each question having five response options scored between 1 and 5. The total score is obtained by summing up the individual scores and dividing the result by the number of questions. A higher score on this scale indicates more severe symptoms. Similarly, the BFCS consists of 8 questions assessing functional capacity, with each question also having five response options scored between 1 and 5. The total score is obtained by summing up the individual scores and dividing the result by the number of questions. A higher score on this scale indicates decreased functional capacity. It is important to note that the questionnaire has been validated and tested for use in the Turkish population.

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Dr. Cemil Taşcıoğlu City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Falsetti P, Conticini E, Baldi C, D'Ignazio E, Al Khayyat SG, Bardelli M, Gentileschi S, D'Alessandro R, D'Alessandro M, Acciai C, Ginanneschi F, Cantarini L, Frediani B. A Novel Ultrasonographic Anthropometric-Independent Measurement of Median Nerve Swelling in Carpal Tunnel Syndrome: The "Nerve/Tendon Ratio" (NTR). Diagnostics (Basel). 2022 Oct 28;12(11):2621. doi: 10.3390/diagnostics12112621. PMID 36359465